CLINICAL TRIAL: NCT02872857
Title: A Pilot Parallel Double-Blind, Randomized Trial of Galantamine for Subarachnoid Hemorrhage
Brief Title: Subarachnoid Hemorrhage Recovery And Galantamine
Acronym: SAHRANG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, HuiMahn Alex Choi, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-16-0228
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Results first posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 8mg galantamine twice daily (Experimental)
  Interventions: Drug: 8mg galantamine twice daily
- 12mg galantamine twice daily (Experimental)
  Interventions: Drug: 12mg galantamine twice daily

INTERVENTIONS:
Drug: Placebo — Placebo will match drug capsules.
  Arms: Placebo
Drug: 8mg galantamine twice daily — Drug will be administered within 36 hours of hospitalization and continued for 90 days.
  Arms: 8mg galantamine twice daily
Drug: 12mg galantamine twice daily — Drug will be administered within 36 hours of hospitalization and continued for 90 days.
  Arms: 12mg galantamine twice daily

SUMMARY:
The purpose of this study is to examine the effects of the study drug--Galantamine-on patients with subarachnoid hemorrhage (SAH). The study will examine how patients with SAH will tolerate the study drug and how it may improve brain functioning in patients after SAH.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous subarachnoid hemorrhage
* Presentation to hospital within 72 hours of symptoms
* Fisher grade 3 hemorrhage (thick subarachnoid clot) on initial computed tomography (CT) scan
* Hunt and Hess grade 1-5 at time of randomization
* Presence of a cerebral aneurysm on computed tomographic angiography (CTA) or Angiogram for which clipping or coiling is possible
* Ability to obtain medication within 36 hours of presentation

Exclusion Criteria:

* subarachnoid hemorrhage (SAH) due to causes other than aneurysm rupture (trauma, arteriovenous malformation (AVM), mycotic aneurysms, Moyamoya)
* Pre-existing disability with modified Rankin Scale (mRS) score ≥2,
* Renal disease as defined by creatinine clearance less than 9 milliliters/min
* History of severe hepatic impairment (Child-Pugh score of 10-15)
* History of chronic obstructive pulmonary disease (COPD) or asthma
* History of dementia
* Co-morbid conditions likely to complicate therapy, including clinically significant arrhythmia, acquired immune deficiency syndrome (AIDS), autoimmune disease, malignancy, and expected mortality within 72 hours
* Expected mortality within 72 hours as determined by PI, treating neurointensivist and neurosurgeon. (Clinically manifested by no attempt at securing aneurysm)
* Females who are pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09; Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huimahn Choi, MD, MS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Houston Methodist Hospital Texas Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Galantamine 8mg During Phase 1: 8mg galantamine twice daily: Drug will be administered within 36 hours of hospitalization and continued for 90 days.
- Placebo During Phase 1; Placebo During Phase 2: Placebo: Placebo will match drug capsules.
- Galantamine 12mg During Phase 2: 12mg galantamine twice daily: Drug will be administered within 36 hours of hospitalization and continued for 90 days.
Period: Phase 1
Arm/Group | Galantamine 8mg During Phase 1 | Placebo During Phase 1 | Galantamine 12mg During Phase 2 | Placebo During Phase 2
Started | 15 | 15 | 0 | 0
Completed | 15 | 15 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Galantamine 8mg During Phase 1 | Placebo During Phase 1 | Galantamine 12mg During Phase 2 | Placebo During Phase 2
Started | 0 | 0 | 15 | 15
Completed | 0 | 0 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Because of the small sample size of this study, which is underpowered to detect differences between the 8mg and 12mg galantamine arms, the pre-specified analysis approach was to combine data for the two galantamine arms when comparing to the placebo arm.
Groups:
- Galantamine: 8mg or 12mg galantamine twice daily: Drug will be administered within 36 hours of hospitalization and continued for 90 days.
- Total: Total of all reporting groups
Arm/Group | Galantamine | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (12.6) | 54.2 (10.4) | 51.25 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 16 | 33
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Tolerability as Assessed by the Number of Participants Who Stop Study Medication Due to Adverse Event Possibly Associated With Study Drug
Time Frame: 90 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 30 | 30
Participants | 1 | 1

2. Primary Outcome: Mortality
Time Frame: 90 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 30 | 30
Participants | 1 | 4

3. Primary Outcome: Modified Rankin Score
Description: The Modified Rankin Score (mRS) is scored as follows:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: 90 days
Population: Data was not collected for 3 in the galantamine arm and 2 in the placebo arm. Because of the small sample size of this study, which is underpowered to detect differences between the 8mg and 12mg galantamine arms, the pre-specified analysis approach was to combine data for the two galantamine arms when comparing to the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 27 | 28
Participants
  0 | 3 | 2
  1 | 8 | 2
  2 | 4 | 12
  3 | 3 | 3
  4 | 4 | 2
  5 | 4 | 3
  6 | 1 | 4

4. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: MoCA scores range between 0 and 30. Higher scores indicate a better outcome, and a score of 26 or over is considered to be normal.
Time Frame: baseline (in hospital)
Population: Data was not collected for 1 in the galantamine arm and 6 in the placebo arm. Because of the small sample size of this study, which is underpowered to detect differences between the 8mg and 12mg galantamine arms, the pre-specified analysis approach was to combine data for the two galantamine arms when comparing to the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 29 | 24
score on a scale | 7.5 (9.2) | 8.2 (8.9)

5. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: as for outcome 4
Time Frame: 90 days
Population: Data was not collected for 6 in the galantamine arm and 6 in the placebo arm. Because of the small sample size of this study, which is underpowered to detect differences between the 8mg and 12mg galantamine arms, the pre-specified analysis approach was to combine data for the two galantamine arms when comparing to the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale | 14.0 (11.5) | 15.8 (10.1)

6. Secondary Outcome: EuroQOL Score as Assessed by a Visual Analogue Scale (VAS)
Description: In the EuroQOL VAS assessment, health status is marked on a 20 cm vertical scale with end points of 0 and 100. 0 corresponds to " the worst health you can imagine," and 100 corresponds to "the best health you can imagine."
Time Frame: 90 days
Population: Data was not collected for 5 in the galantamine arm and 6 in the placebo arm. Because of the small sample size of this study, which is underpowered to detect differences between the 8mg and 12mg galantamine arms, the pre-specified analysis approach was to combine data for the two galantamine arms when comparing to the placebo arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 25 | 24
units on a scale | 76.2 (19.4) | 74.0 (22.6)

ADVERSE EVENTS:
Time Frame: 90 days
Description: Because of the small sample size of this study, which is underpowered to detect differences between the 8mg and 12mg galantamine arms, the pre-specified analysis approach was to combine data for the two galantamine arms when comparing to the placebo arm.
Arm/Group | Galantamine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/30 | 4/30
Serious Adverse Events (participants affected / at risk) | 17/30 | 17/30
Other Adverse Events (participants affected / at risk) | 26/30 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine (N=30) | Placebo (N=30)
Delayed Cerebral Ischemia (Vascular disorders) | 10 (12) | 12 (15)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Cerebral Edema (Nervous system disorders) | 3 (3) | 3 (3)
Clinical Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 2 (2)
Angio Complication (Vascular disorders) | 1 (1) | 1 (1)
Surgical Complication (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine (N=30) | Placebo (N=30)
Anemia (Blood and lymphatic system disorders) | 13 (13) | 12 (12)
Hyponatremia (Metabolism and nutrition disorders) | 12 (12) | 11 (12)
Bradycardia (Cardiac disorders) | 10 (10) | 12 (12)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 6 (6)
Hypernatremia (Metabolism and nutrition disorders) | 7 (7) | 11 (11)
Univary Tract Infections (Renal and urinary disorders) | 9 (9) | 5 (5)
Tachycardia (Cardiac disorders) | 8 (8) | 5 (5)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 5 (5)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1)
Angio Complication (Vascular disorders) | 1 (2) | 0 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Nausea (General disorders) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Other (General disorders) | 20 (36) | 16 (39)
Clinical Seizure (Nervous system disorders) | 1 (2) | 2 (2)
Pulmonary Edema (Cardiac disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT02872857/Prot_SAP_000.pdf